CLINICAL TRIAL: NCT00353587
Title: Phase 2/3, Randomized, Double-blind, Placebo- and Active Comparator-controlled, Parallel, Multicenter Study to Determine Safety and Efficacy of Metaglidasen in Treatment of Type 2 Diabetes Suboptimally Controlled on Insulin
Brief Title: Safety and Efficacy Study of Metaglidasen in Type 2 Diabetes in Patients Suboptimally Controlled on Insulin
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M102-20509
Record Dates: First submitted 2006-07-14; First posted 2006-07-18 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Type 2 Diabetes
Keywords: insulin sensitizer; type 2 diabetes; diabetes; glucose control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — arhalofenate; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- MBX-102 200 mg (Experimental): MBX-102 200 mg once daily for 16 weeks
  Interventions: Drug: MBX-102
- MBX-102 400 mg (Experimental): MBX-102 400 mg once daily for 16 weeks
  Interventions: Drug: MBX-102
- MBX-102 600 mg (Experimental): MBX-102 600 mg once daily for 16 weeks
  Interventions: Drug: MBX-102
- Sugar Pill (Placebo Comparator): Placebo comparator once daily for 16 weeks
  Interventions: Drug: Placebo
- Actos (Active Comparator): Actos 30 mg once daily for 16 weeks
  Interventions: Drug: Actos

INTERVENTIONS:
Drug: MBX-102 — MBX-102 200 mg once daily for 16 weeks
  Arms: MBX-102 200 mg
Drug: MBX-102 — MBX-102 400 mg once daily for 16 weeks
  Arms: MBX-102 400 mg
Drug: MBX-102 — MBX-102 600 mg once daily for 16 weeks
  Arms: MBX-102 600 mg
Drug: Placebo — MBX-102 Placebo once daily for 16 weeks
  Arms: Sugar Pill
Drug: Actos — Actos 30 mg once daily for 16 weeks
  Arms: Actos

SUMMARY:
This is a multicenter, randomized, double-blind, placebo- and active comparator-controlled phase 2/3 study of three dose levels of MBX-102 (200, 400, 600 mg) given orally to patients with type 2 diabetes receiving concomitant therapy with insulin. Eligible patients will be adults with type 2 diabetes who are taking intermediate- and/or long-acting insulin or pre-mixed (e.g., "70/30") insulin, or a combination of insulin and one or two non-TZD hypoglycemic agents including sulfonylurea, metformin, acrabose or Byetta, but who are poorly controlled on their existing therapy. Preference for enrollment will be given to patients on insulin monotherapy. Patients treated with a combination of insulin and other hypoglycemic agent(s) must be willing and able to discontinue and washout of the hypoglycemic agent(s) for the entire duration of the study (in toto, approximately 28 weeks). Patients who are taking fixed doses of a short-acting insulin (e.g., not a "sliding scale") in combination with intermediate-acting insulin may qualify for the study if both the patient and investigator are willing to either change to pre-mixed insulin (e.g., 70/30) or discontinue use of the short acting insulin for at least 26 weeks. Patients treated with a sliding scale of short-acting insulin will not be eligible for enrollment.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo- and active comparator-controlled phase 2/3 study of three dose levels of MBX-102 (200, 400, 600 mg) given orally to patients with type 2 diabetes receiving concomitant therapy with insulin. Eligible patients will be adults with type 2 diabetes who are taking intermediate- and/or long-acting insulin or pre-mixed (e.g., "70/30") insulin, or a combination of insulin and one or two non-TZD hypoglycemic agents including sulfonylurea, metformin, acrabose or Byetta, but who are poorly controlled on their existing therapy. Preference for enrollment will be given to patients on insulin monotherapy. Patients treated with a combination of insulin and other hypoglycemic agent(s) must be willing and able to discontinue and washout of the hypoglycemic agent(s) for the entire duration of the study (in toto, approximately 28 weeks). Patients who are taking fixed doses of a short-acting insulin (e.g., not a "sliding scale") in combination with intermediate-acting insulin may qualify for the study if both the patient and investigator are willing to either change to pre-mixed insulin (e.g., 70/30) or discontinue use of the short acting insulin for at least 26 weeks. Patients treated with a sliding scale of short-acting insulin will not be eligible for enrollment.

Following any insulin dose adjustment during the first few weeks of the study, insulin dose and regimen should remain constant for the duration of the study.

No stand alone (e.g., other than pre-mixed) short- or ultrashort-acting insulin and/or sliding scale will be allowed for the entire duration of the study.

A minimum of 400 patients will be randomized in this study (approximately 80 to each of the five treatment arms). Additional patients may be enrolled as appropriate to replace screen failures and drop-outs during the initial period of the study.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes (as described by the Expert Committee on the Diagnosis and Classification of Diabetes Mellitus24) treated with insulin alone (a stable dose of long and/or intermediate-acting insulin or pre-mixed insulin e.g., "70/30") ≥ 30 units/day for at least 3 months, but poorly controlled on their existing therapy
* Or, patients treated with insulin (as above) in combination with non-TZD hypoglycemic agents (e.g., a sulfonylurea, metformin, acrabose, or Byetta for at least 3 months, but poorly controlled on their existing therapy
* Or, patients treated with fixed doses of short-acting insulin in combination with intermediate-acting insulin for at least 3 months, but poorly controlled on their existing therapy
* Patients in last 2 categories must be willing to discontinue the use of OHA and/or short-acting insulin (or change to pre-mixed insulin) for at least 26 weeks.
* Male or female, 18-75 years of age
* Provide informed consent and agree to comply with study requirements
* Current monotherapy insulin dose regimen ≥ 30 units/day (stable for 8-week Run-in/stabilization Period); or patients who need insulin dose adjustment must have a stabilized dose ≥ 30 units/day. Patients must not have taken TZDs within 5 months of screening
* All female patients must be surgically sterile, post-menopausal (at least 40 years of age with no history of menses for at least 2 years) or agree to use adequate contraception(s) that must include a barrier method (other methods may include oral contraceptives, double barrier methods, intra-uterine devices, or abstinence). Depo contraceptives are excluded
* Female patients must not be pregnant or lactating
* BMI 26-44 kg/m2
* Hemoglobin A1c must be ≥7.5%, ≤11.5% at both Screening and Visit 4
* Patients must have a FPG ≤ 220 mg/dl
* Patients must have liver function tests ≤ 2X the upper limits of normal for AST, ALT, and bilirubin, and ≤ 2.5X the upper limits of normal for ALP and GGT
* Patients must have serum creatinine ≤ 1.8 mg/dl for males and ≤ 1.5 mg/dl for females and BUN ≤ 40 mg/dl
* Fecal occult blood test must be negative
* All other clinical laboratory parameters must be within normal limits or considered not clinically significant for participation in this study, including: hematology, coagulation, other serum chemistry, and other urinalysis parameters
* TSH must be ≤ 3x ULN and patient clinically euthyroid in opinion of investigator. If TSH is > ULN but ≤ 3x ULN, and patient is clinically euthyroid, FT4 should be drawn and must be WNL
* Electrocardiogram (ECG) must be normal, or considered not clinically significant, for participation in this study
* Patients must have a blood pressure ≤ 160/90 mm/hg including hypertensive patients controlled with medication

Exclusion Criteria:

Patients will be excluded from study participation if any of the following applies:

* History of diabetes secondary to pancreatitis or pancreatectomy
* Requirement for short-acting insulin during the study
* Weight loss > 10 pounds in the three months prior to study
* History of TZD use (Actos or Avandia) within 5 months of Screening Visit
* History of TZD discontinuation due to side effect or lack of efficacy
* Prior history of endoscopically or radiographically documented peptic ulcer disease within last 5 years (unless patient had documented H. pylori infection with subsequent treatment and no recurrence)
* Prior history of GI bleeding within last 5 years (except for hemorrhoids or perianal disease)
* Known infection with the human immunodeficiency virus (HIV) or history of viral hepatitis type B or C
* History of congestive heart failure within last 5 years (NYHA Class III-IV)
* History of significant pulmonary disease, myocardial infarction, cerebrovascular accident, or nephrotic syndrome within last 1 year
* Elevated creatine phosphokinase (> 2X the upper limits of normal)
* Malignancy within the last 5 years (except resected basal cell carcinoma)
* Ongoing active infection, as evidenced by symptoms such as temperature > 38.5° C and/or clinically significant elevation in WBC count (i.e., not asymptomatic colonization)
* Change in treatment with lipid-lowering agent after screening visit
* Current or expected requirement for anticoagulant therapy [except for low- dose (≤ 325 mg/d) aspirin]
* Current or expected treatment with phenytoin
* Current or anticipated treatment with non-steroidal anti-inflammatory drugs (i.e., naproxen, ibuprofen, Vioxx, Celebrex, indomethacin, etc.). However, patients may take aspirin < 325 mg/day for cardiovascular prophylaxis
* Known hypersensitivity to NSAIDs
* Treatment with any other investigational therapy within the 30 days prior to Screening Visit
* History of illicit drug or alcohol abuse within last 1 year
* Current or expected treatment with systemic corticosteroids (except topical, ophthalmic, intra-articular, or inhaled at a dose < 1600 μg/day)
* Any other condition that compromises the ability of the patient to provide informed consent or to comply with the objectives and procedures of this protocol, as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2006-05; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Evaluate effects of MBX-102 administered orally at doses of 200, 400 and 600 mg daily for 16 weeks, on glucose control, as measured by HbA1c
Evaluate safety of MBX-102 with particular emphasis on endpoints of weight gain and edema

CONTACTS AND LOCATIONS:
Locations (67):
- United States (18):
  - NEA Clinic, Jonesboro, Arkansas
  - Associated Pharmaceutical Research Center, Inc., Buena Park, California
  - The Intermed Group, Los Angeles, California
  - LAC/USC Medical Center, Los Angeles, California
  - International Research Associates, LLC, Miami, Florida
  - Suncoast Clinical Research, Inc., Palm Harbor, Florida
  - Andres Patron DO PA, Pembroke Pines, Florida
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Clinical Investigation Specialists, Inc., Gurnee, Illinois
  - Olive Branch Research, Olive Branch, Mississippi
  - Optimed Research, LLC, Columbus, Ohio
  - Radiant Research - Greer, Greer, South Carolina
  - Dallas Diabetes & Endocrine Center, Dallas, Texas
  - Mercury Pharma Services, Houston, Texas
  - Diabetes Center of the Southwest, Midland, Texas
  - Diabetes & Glandular Disease Research Associates, P.A., San Antonio, Texas
  - McGuire VA Medical Center, Richmond, Virginia
  - National Clinical Research, Richmond, Virginia
- Argentina (17):
  - Consultorio Integral de Atencion al Diabetico (CIAD), Buenos Aires
  - CIMEL, Buenos Aires
  - Centro de Atencion Integral en Diabetes, Endocrinologica y Metabolismo, Buenos Aires
  - Fundacion CIDEA, Buenos Aires
  - Sanatorio Municipal Dr. Julio Mendez, Buenos Aires
  - Instituto Medico Especializado, Buenos Aires
  - Hospital Thompson, Buenos Aires
  - Clinica Dleta Zarate, Buenos Aires
  - Hospital Privado de Comunidad, Buenos Aires
  - Consultorios Asociados de Endocrinologia, Capital Federal
  - Instituto Latinoamericano de Investigaciones Clinicas, Córdoba
  - Sanatorio Parque, Córdoba
  - Fundacion Marcelino Rusculleda Batlle, Córdoba
  - Instituto de Clinica Medica y Diabetes, Mendoza
  - Policlio Modelo de Cipoletti, Rio Negro
  - Hospital San Bernardo, Salta
  - CER San Juan Centro Polivalente de Asistencia e Investigacion Clinica, San Juan Capital
- India (18):
  - Nizam's Institute of Medical Sciences, Panjagutta, Hyderabad, Andhra Pradesh
  - Bharti Research Institute of Diabetes & Endocrinology, Karnāl, Haryana
  - Amrita Institute of Medical Sciences, Kochi, Kerala
  - Kasturba Medical College Hospital, Attavar, Mangalore
  - Sterling Hospital, Ahmedabad
  - St. John's Medical College Hospital, Bangalore
  - M.S. Ramaih Medical College & Hospital, Bangalore
  - Diacon Hospital, Bangalore
  - Sri Ramachandra Medical Centre, Chennai
  - Dr. V. Seshiah Diabetes Care & Research Institute, Chennai
  - Apollo Gleneages/Dept. of Endocrinology, Kolkata
  - Diabetes Care and Research Center, Maharashtra
  - Kasturba Hospital, Manipal
  - Chowpatty Medical Center, Mumbai
  - Mediheights Healthcare Pvt. Ltd., Mumbai
  - KEM Hospital, Pune
  - Kerala Institute of Medical Sciences, Trivandrum
  - Christian Medical College Hospital, Vellore
- Israel (14):
  - Endocrinology Institute, Haemek Medical Center, Afula
  - Barzilai Medical Center, Ashkelon
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Linn Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Hadassah University Hospital, Jerusalem
  - Clalit Health Services, Jerusalem
  - Institution of Diabetes and Metabolism, Nahariya
  - Endocrinology & Diabetes Institute, Petah Tikva
  - Department of Endocrinology, Ziv Medical Center, Safed
  - Zamenhoff Medical Center, Tel Aviv
  - Institute of Metabolic Diseases, Tel Aviv
  - Assaf Haroffe Medical Center, Zrifin